CLINICAL TRIAL: NCT05808894
Title: Extended Pancreatic Neck Transection Versus Conventional Pancreatic Neck Transection During Laparoscopic Pancreaticoduodenectomy( LPDEXCEPT): a Multicenter Randomized Controlled Trial
Brief Title: Extended Pancreatic Neck Transection Versus Conventional Pancreatic Neck Transection During Laparoscopic Pancreaticoduodenectomy( LPDEXCEPT)
Acronym: LPDEXCEPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinrui Zhu，MD (Other)
Collaborators: The Affiliated Hospital Of Guizhou Medical University (Other); Shandong Provincial Hospital (Other Government); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Xinrui Zhu，MD, attending doctor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-167-1
Record Dates: First submitted 2023-03-14; First posted 2023-04-12 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Laparoscopic Pancreaticoduodenectomy
Keywords: laparoscopic pancreaticoduodenectomy; pancreatic neck transection level

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extended transection group (Experimental): the patients in extended transection group obtain extended pancreatic neck transection during laparoscopic pancreaticoduodenectomy.
  Interventions: Procedure: extended pancreatic neck transection during laparoscopic pancreaticoduodenectomy
- conventional transection group (No Intervention): the patients in conventional transection group obtain conventional pancreatic neck transection during laparoscopic pancreaticoduodenectomy.

INTERVENTIONS:
Procedure: extended pancreatic neck transection during laparoscopic pancreaticoduodenectomy — Transect the pancreatic neck at ≥5mm and ≤10mm beyond the left side of the portal vein.
  Arms: extended transection group

SUMMARY:
The investigators conduct the clinical randomized controlled trial to evaluate the superiority of extended pancreatic neck transection during laparoscopic pancreaticoduodenectomy (LPD). The participants in the study group obtain extended pancreatic neck transection during LPD, while participants in the control group conventional pancreatic neck transection. The purposes of this study include: 1.Primary objective: To compare the incidence of clinically relevant pancreatic fistula (grades B-C according International Study Group on Pancreatic Surgery) between the study group and the control group. 2.Secondary objective: To compare the incidence of postoperative morbidity (Clavien-Dindo score ≥3）between the two groups. To compare the location of pancreatic duct and the surgical performance of pancreaticojejunostomy between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with benign or resectable malignant tumors of the lower common bile duct, Vater ampulla, head or uncinate process of the pancreas.
2. 18 years old < age < 80 years old, no gender limit.
3. Patient is expected survival beyond 3 months.
4. No pregnancy or pregnancy plan within 3 months after surgery.
5. Nutrition risk score <3 according to the Nutritional Risk Screening for Inpatients 2002 (NRS2002) standard score.
6. No contraindication to surgery for anesthetic evaluation.
7. The subjects voluntarily joined the study and signed an informed consent form, with good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Patients with borderline resectable and unresectable malignancies.
2. Patients undergoing neoadjuvant chemotherapy or radiotherapy.
3. Patients with tumors exceeding the level of the gastroduodenal artery as measured by preoperative radiography.
4. Intraoperative exploration reveals tumor adhesions with portal vein-superior mesenteric vein, requiring revascularization and reconstruction.
5. Operation transfers to open.
6. Operation transfers to other procedure.
7. The main pancreatic duct can not be found intraoperatively, the duct-to-mucosa pancreaticojejunostomy can not be operated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
the incidence of clinically relevant pancreatic fistula | 3 months postoperatively
  the incidence of the clinically relevant pancreatic fistula according the International Study Group of Pancreatic Surgery's definition and grading

SECONDARY OUTCOMES:
location of the pancreatic duct in the pancreatic transverse section | intraoperatively
  Before performing the pancreaticojejunostomy, place the pancreatic transverse section in the central position of the lens. Measure the anterior-posterior diameter of the pancreas and the distance of the pancreatic duct from the back of the pancreas. The location of the pancreatic duct in the pancreatic transverse section is equal to the ratio of the distance of the pancreatic duct from the back of the pancreas to the anterior-posterior diameter of the pancreas.
surgical performance of pancreaticojejunostomy | intraoperatively
  the duration of pancreaticojejunostomy
postoperative morbidity | 3 months postoperatively
  postoperative morbidity (Clavien-Dindo score ≥3）within 3 months postoperatively
postoperative mortality | 3 months postoperatively
  mortality within 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Bing Peng, Professor, Study Chair — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardol T, Delicque J, Hermida M, Herrero A, Guiu B, Fabre JM, Souche R. Neck transection level and postoperative pancreatic fistula after pancreaticoduodenectomy: A retrospective cohort study of 195 patients. Int J Surg. 2020 Oct;82:43-50. doi: 10.1016/j.ijsu.2020.08.001. Epub 2020 Aug 22. PMID 32841726
- [Background] Jwa EK, Hwang S. Extended pancreatic transection for secure pancreatic reconstruction during pancreaticoduodenectomy. Ann Hepatobiliary Pancreat Surg. 2017 Aug;21(3):138-145. doi: 10.14701/ahbps.2017.21.3.138. Epub 2017 Aug 31. PMID 28990000
- [Background] Strasberg SM, Drebin JA, Mokadam NA, Green DW, Jones KL, Ehlers JP, Linehan D. Prospective trial of a blood supply-based technique of pancreaticojejunostomy: effect on anastomotic failure in the Whipple procedure. J Am Coll Surg. 2002 Jun;194(6):746-58; discussion 759-60. doi: 10.1016/s1072-7515(02)01202-4. PMID 12081065
- [Background] Subar D, Pietrasz D, Fuks D, Gayet B. A novel technique for reducing pancreatic fistulas after pancreaticojejunostomy. J Surg Case Rep. 2015 Jul 9;2015(7):rjv074. doi: 10.1093/jscr/rjv074. PMID 26160766
- [Derived] You J, Zhang J, Cai H, Wang X, Wang H, Li Y, Yu C, Wang L, Zhou X, Peng B, Cai Y. Extended pancreatic neck transection versus conventional pancreatic neck transection during laparoscopic pancreaticoduodenectomy (LPDEXCEPT): protocol for a multicentre superiority randomised controlled trial. BMJ Open. 2024 Jan 10;14(1):e078092. doi: 10.1136/bmjopen-2023-078092. PMID 38199635